CLINICAL TRIAL: NCT06975995
Title: A Postbiotics Improves the Quality of Life and Nutritional Status in Elderly Hemodialysis Patients
Brief Title: Effect of the Postbiotics on Complications Treatment in Elderly Hemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Bio-EHD
Record Dates: First submitted 2024-06-02; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-06

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group will receive oral postbiotics product for 150ml per day during the treatment period (from week 1 to week 12). Then, the group will end the trial.
  Interventions: Dietary Supplement: Yi'en Yuan Honey Fermented Drink
- Placebo group (Placebo Comparator): The placebo group will receive oral placebo during the treatment period (from week 1 to week 12). Then, the group will enter into remedial the treatment period (from week 13 to week 24) and receive the same oral postbiotics product as intervention group for 150ml per day. The group will end the trial at week 24.
  Interventions: Dietary Supplement: Yi'en Yuan Honey Fermented Drink

INTERVENTIONS:
Dietary Supplement: Yi'en Yuan Honey Fermented Drink — The oral postbiotics product used in the trial is called Yi'en Yuan Honey Fermented Drink. The product is made from water, edible brown sugar, and honey as raw materials. It is fermented by a mixture of plant lactic acid bacteria and coagulating Bacillus, and then inactivated at high temperature. The product meets the food and beverage standard. Participants will receive the product for 150ml per day.

SUMMARY:
The purpose of the trial is to explore the effect of exogenous postbiotics supply on the quality of life and nutritional status of elderly hemodialysis patients.

Participants will be devided into intervention group and placebo group in an 1:1 ratio.They will:

1. In the treatment period for 12 weeks, intervention group receives postbiotics product while the other group receives placebo.
2. In the subsequent 12 weeks, intervention group ends the trial and placebo group enters into remedial treatment period. Placebo group will receive postbiotics product for 12 weeks.

Researchers will analyze the change of indicators such as quality of life and nutrition state of participants from the baseline to end of treatment, and compare the difference between the two group.

DETAILED DESCRIPTION:
Intestinal flora imbalance has a high prevalence in CKD patients and is closely invloved with CKD complications like malnutrition and anemia, which affects quality of life and long-term prognosis of CKD patients. Probiotics is the bioactive compound produced by probiotics when it consumes prebiotics. It can alleviate the condition and improve quality of life of patients by regulating growth of microbiota directly and indirectly and inhibiting growth of pathogenic microorganism. The purpose of the trial is to explore the effect of exogenous postbiotics supply on the quality of life and nutritional status of elderly hemodialysis patients.

The study is a multicenter prospective open-labled and randomized controlled trial. Elderly patients with age ≥65 years and received hemodialysis treatment for more than 6 months will be included in the study. During the screen period, the patients with medical history that might affect oral feeding or gastrointestinal functions will be excluded.

After enrollment, the patients will be educated about how to keep diet records and then they will be randomly divided into group A (intervention group) and group B (placebo group) in an 1:1 ratio. The patients in group A will receive oral postbiotics and group B receive placebo. The treatment period is 12 weeks. Subsequently, group A ends the trial, and group B enters the remedial treatment period, receiving oral postbiotics, and the treatment cycle is 12 weeks.

At 0, 12 and 24 weeks quality of life score, nutrition evaluation, diet status and gastrointestinal symptom score respectively will be evaluated. The stool and serum of patients will be collected for intestinal flora and urotoxins measurements. Besides, the trial will collect routine biochemical indicators. The investigators will analyze those indicators above from the baseline to end of treatment and compare the difference between intervention group and placebo group.

ELIGIBILITY:
Inclusion Criteria:

Investigators must maintain a screening log of all potential study candidates that includes limited information about the potential candidate, date, and outcome of the screening process (e.g. enrolled into study, reason for ineligibility, or refused to participate). After signing an informed consent form, potential patients must meet all of the criteria:

1. Age ≥65 years.
2. Receiving maintenance hemodialysis therapy for at least 6 months.

Exclusion Criteria:

The following exclusion criteria must NOT be present for each subject:

1. Subjects with medical history that might affect oral feeding (e.g. intestinal obstruction, gastrointestinal bleeding, acute pancreatitis and accidental inhalation) within the last 1 month prior to screening.
2. Subjects with medical history that might affect gastrointestinal functions (e.g. inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), short bowel syndrome (SBS), et al.).
3. Subjects who cannot communicate and collaborate normally.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes of nutritional status from the baseline to the 12th week of treatment period and differences between the intervention group and the placebo group. | baseline, the 12th week of treatment period
  Nutritional status of the patient is defined as the results of physical examination and SGA-7 rating scale.
Changes of gastrointestinal symptoms from the baseline to the 12th week of treatment period and differences between the intervention group and the placebo group. | baseline, the 12th week of treatment period
  Gastrointestinal symptoms of the patient is defined as the scores of gastrointestinal symptom rating scale (GSRS).
Changes of quality of life from the baseline to the 12th week of treatment period and differences between the intervention group and the placebo group. | baseline, the 12th week of treatment period
  Quality of life of the patient is defined as the scores of kidney disease life quality scale (SF-36) .
Changes of asthenia of the patients from the baseline to the 12th week of treatment period and differences between the intervention group and the placebo group. | baseline, the 12th week of treatment period
  Asthenia of the patients is defined as the scores of edmonton frail Scale (EFS).
Changes of body mass index from the baseline to the 12th week of treatment period and differences between the intervention group and the placebo group. | baseline, the 12th week of treatment period
  The BMI (kg/m2) of the patients.
Changes of dry weight from the baseline to the 12th week of treatment period and differences between the intervention group and the placebo group. | baseline, the 12th week of treatment period
  The dry weight of the patient is obtained from the bioelectrical impedance analysis.

SECONDARY OUTCOMES:
Changes of IS level from baseline to the end of treatment and difference between the intervention and placebo group. | baseline, the 12th week of treatment period
  Enterogenous urotoxin level is defined as the serum level of IS. The levels of serum IS will be measured by mass spectrometry.
Changes of TMAO level from baseline to the end of treatment and difference between the intervention and placebo group. | baseline, the 12th week of treatment period
  Enterogenous urotoxin level is defined as the serum level of TMAO. The levels of serum TMAO will be measured by mass spectrometry.
Changes of PCS level from baseline to the end of treatment and difference between the intervention and placebo group. | baseline, the 12th week of treatment period
  Enterogenous urotoxin level is defined as the serum level of PCS. The levels of serum PCS will be measured by mass spectrometry.
Changes of hemoglobin from the baseline to the end of treatment, and differences between the intervention group and the placebo group. | baseline, the 12th week of treatment period
  The levels of hemogolbin (g/L).
Changes of albumin from the baseline to the end of treatment, and differences between the intervention group and the placebo group. | baseline, the 12th week of treatment period
  The levels of albumin (g/L)
Changes of BUN from the baseline to the end of treatment, and differences between the intervention group and the placebo group. | baseline, the 12th week of treatment period
  The levels of BUN (mmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Chen, Study Chair — Peking University First Hospital
Locations (1):
- Peking UFH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data of participants of the study will keep confidential and there is no plan to share IPD to other researchers.

DOCUMENTS (1):
  • Study Protocol (2023-05-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT06975995/Prot_000.pdf